CLINICAL TRIAL: NCT03401879
Title: Retinal Neuro-vascular Coupling in Patients With Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Section Head Ophthalmo-Pharmacology, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-210417
Record Dates: First submitted 2018-01-10; First posted 2018-01-17 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Optic Neuritis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Optic Neuritis | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with MS (Experimental): Patients with Multiple Sclerosis
  Interventions: Device: Dynamic Vessel Analyzer (DVA); Device: Fourier Domain Doppler Optical Coherence Tomography (FDOCT); Device: Optical coherence tomography (OCT); Device: Optical coherence tomography angiography (OCTA)
- Healthy control subjects (Experimental): Healthy age- and sex- matched control subjects
  Interventions: Device: Dynamic Vessel Analyzer (DVA); Device: Fourier Domain Doppler Optical Coherence Tomography (FDOCT); Device: Optical coherence tomography (OCT); Device: Optical coherence tomography angiography (OCTA)

INTERVENTIONS:
Device: Dynamic Vessel Analyzer (DVA) — Retinal vessel diameters and oxygen saturation will be measured with the DVA device.
Device: Fourier Domain Doppler Optical Coherence Tomography (FDOCT) — Retinal blood flow will be assessed using FDOCT.
Device: Optical coherence tomography (OCT) — Nerve fiber layer thickness and central retinal thickness will be measured using OCT.
Device: Optical coherence tomography angiography (OCTA) — Retinal microvasculature will be assessed using OCTA.

SUMMARY:
Multiple sclerosis (MS) affects approximately 2.3 million patients worldwide, with a global median prevalence of 33 per 100,000. MS is diagnosed at an average of 30 years and affects twice as many women as men. MS is traditionally diagnosed by the presentation of lesions of the central nervous system, disseminated in time and in space, proven by clinical examination and magnetic resonance imaging. Several anatomical parameters in the eye, both vascular and neural, have been found to be altered in MS patients.

Because of its unique optical properties, the eye offers the possibility of the non-invasive assessment of both structural and functional alterations in neuronal tissue. As the neuro-retina is part of the brain, it does not come as a surprise that neuro-degenerative changes in the brain are accompanied by structural and possibly also functional changes in the neuro-retina and the ocular vasculature.

The current study seeks to test the hypothesis that beside the known anatomical changes, also functional changes can be detected in the retina of patients with MS. For this purpose, flicker light induced hyperemia will be measured in the retina as a functional test to assess the coupling between neural activity and blood flow. Further, structural parameters such as retinal nerve fiber layer thickness and function parameters such as ocular blood flow and retinal oxygenation will be assessed and compared to age and sex matched controls.

ELIGIBILITY:
Inclusion criteria for healthy subjects:

* Men and women aged over 18 years
* Non-smokers
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropy < 6 Dpt.

Inclusion criteria for patients with MS:

* Men and women aged over 18 years
* Diagnosis of relapsing-remitting multiple sclerosis (RRMS) according to clinical evaluation and McDonald criteria (revision 2010)
* History of AON in one eye at least one year ago
* Non-smokers
* Normal ophthalmic findings, ametropy < 6 Dpt.
* Adequate visual acuity to allow participation in the ocular blood flow measurements
* A potential participant has to be on stable doses of all medications he/she is taking because of consisting illnesses according to medical history (except MS therapy itself which will be recorded separately) for at least 30 days prior inclusion, if considered relevant by the investigator.

Any of the following will exclude a healthy subject from the study:

* Diagnosis of "possible MS" according to the McDonald criteria (revision 2010)
* Presence or history of a severe medical condition as judged by the clinical investigator
* Untreated Arterial hypertension
* History or family history of epilepsy
* Presence of any abnormalities preventing reliable measurements in the study eye as judged by the investigator
* Family history of MS, optic neuritis, neuromyelitis optica (NMO, Devic disease) or NMO spectrum disorders
* History of inflammatory or infectious disease of central nervous system
* Best corrected visual acuity < 0.5 Snellen
* Ametropy ≥ 6Dpt
* Pregnancy or planned pregnancy
* Alcoholism or substance abuse

Any of the following will exclude a patient from the study:

* Presence or history of a severe medical condition other than MS as judged by the clinical investigator
* History of neuromyelitis optica (NMO, Devic disease) or NMO spectrum disorders
* History of inflammatory or infectious disease of central nervous system other than MS
* Untreated Arterial hypertension
* History or family history of epilepsy
* Presence of any abnormalities preventing reliable measurements in the study eye as judged by the investigator
* Best corrected visual acuity < 0.5 Snellen
* Ametropy ≥ 6 Dpt
* Pregnancy, planned pregnancy
* Significant neurological disease other than MS, if considered relevant by the investigator
* Alcoholism or substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Flicker induced increase in retinal blood flow | 1 day
  Response of retinal blood flow to flicker light assessed with FDOCT

SECONDARY OUTCOMES:
Retinal vessel diameters | 1 day
  Response of retinal vessel diameters to flicker light assessed with DVA
Retinal oxygen saturation | 1 day
  Retinal oxygen saturation measured with DVA
Retinal nerve fiber layer thickness | 1 day
  Retinal nerve fiber layer thickness measured using OCT
Layer specific flow signal | 1 day
  Retinal layer specific blood flow signal measured using OCTA

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhöfer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria, Austria

REFERENCES:
- [Derived] Kallab M, Hommer N, Schlatter A, Bsteh G, Altmann P, Popa-Cherecheanu A, Pfister M, Werkmeister RM, Schmidl D, Schmetterer L, Garhofer G. Retinal Oxygen Metabolism and Haemodynamics in Patients With Multiple Sclerosis and History of Optic Neuritis. Front Neurosci. 2021 Oct 12;15:761654. doi: 10.3389/fnins.2021.761654. eCollection 2021. PMID 34712117